CLINICAL TRIAL: NCT05147350
Title: Phase 1 Study of the PKMYT1 Inhibitor RP-6306 in Combination With FOLFIRI for the Treatment of Advanced Solid Tumors
Brief Title: Study of RP-6306 With FOLFIRI in Advanced Solid Tumors
Acronym: MINOTAUR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to terminate the study
Sponsor: Debiopharm International SA (Industry)
Collaborators: Repare Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP-6306-03
Record Dates: First submitted 2021-11-03; First posted 2021-12-07 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — IFL protocol

STUDY DESIGN:
Intervention Model Description: Dose Escalation and expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1: RP-6306 in combination with FOLFIRI Dose Escalation (Experimental): RP-6306 will be administered as oral capsules Multiple dose levels of RP-6306 (oral) and FOLFIRI (IV)
  Interventions: Drug: RP-6306 (oral PKMYT1 inhibitor)

INTERVENTIONS:
Drug: RP-6306 (oral PKMYT1 inhibitor) — RP-6306 (Oral) in combination with FOLFIRI (IV)
  Other Names: FOLFIRI

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of RP-6306 with FOLFIRI in patients with eligible advanced solid tumors, determine the maximum tolerated dose (MTD), identify a recommended phase 2 dose (RP2D) and preferred schedule, and assess preliminary anti-tumor activity.

DETAILED DESCRIPTION:
To assess the safety and tolerability of RP-6306 in combination with FOLFIRI in patients with eligible, advanced solid tumors. Incidence and severity of treatment-emergent adverse events (TEAEs), laboratory assessments, vital signs, electrocardiograms (ECGs), and use of concomitant medications.

The Sponsor of the study has changed from 'Repare Therapeutics' to 'Debiopharm International SA' in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and ≥18 years-of-age at the time of signature of the informed consent
* Confirmed advanced solid tumors resistant or refractory to standard treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* All patients must have locally advanced or metastatic CRC, GI, or esophageal cancer(s) and radiographic evidence of progressing disease.
* Measurable disease as per RECIST v1.1
* Submission of available tumor tissue or willingness to have a biopsy performed if safe and feasible
* Acceptable hematologic and organ function at screening
* Negative pregnancy test for women of childbearing potential at Screening and prior to first study drug.

Exclusion Criteria:

* Inability to swallow and retain oral medications.
* Chemotherapy or small molecule antineoplastic agent given within 21 days or <5 half- lives, whichever is shorter, prior to first dose of study treatment.
* History or current condition, therapy, or laboratory abnormality that might confound the study results, or interfere with the patient's participation for the full duration of the study treatment.
* Patients who are pregnant or breastfeeding
* Life-threatening illness, medical condition, active uncontrolled infection, or organ system dysfunction or other reasons which, in the investigator's opinion, could compromise the participating patient's safety.
* Major surgery within 4 weeks prior to first study treatment dose.
* Uncontrolled, symptomatic brain metastases.
* Uncontrolled high blood pressure
* Active, uncontrolled bacterial, fungal, or viral infection, including hepatitis B virus (HBV), hepatitis C virus (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS) related illness.
* Moderate or severe hepatic impairment
* Cardiac diseases currently or within the last 6 months as defined by New York Heart Association (NYHA) ≥Class 2
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - #1019, UCLA, Westwood Cancer Center, Los Angeles, California
  - #1022, Moffitt Cancer Center, Tampa, Florida
  - #1008, Columbia University, New York, New York
  - #1001, The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - #1013, The University of Utah, Huntsman Cancer Center, Salt Lake City, Utah
- # 2001, Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Spain (2):
  - # 5002, South Texas Accelerated Research Therapeutics, Madrid
  - # 5003, Hospital Universitario HM Sanchinarro, Madrid
- # 3003, Sarah Cannon Research Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 40 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI: 40 mg QD oral (PO) lunresertib daily in combination with 180 mg/m2 intravenous (IV) irinotecan given over 30 to 90 minutes, 400 mg/m2 IV leucovorin given over 30 to 90 minutes with irinotecan, and 400 mg/m2 IV fluorouracil bolus after leucovorin, then 2400 mg/m2 IV continuous IV of fluorouracil over 46 hours (Days 1 and 2) of each 14-day cycle
- 120 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI: 120 mg QD oral (PO) lunresertib daily in combination with 180 mg/m2 intravenous (IV) irinotecan given over 30 to 90 minutes, 400 mg/m2 IV leucovorin given over 30 to 90 minutes with irinotecan, and 400 mg/m2 IV fluorouracil bolus after leucovorin, then 2400 mg/m2 IV continuous IV of fluorouracil over 46 hours (Days 1 and 2) of each 14-day cycle
- 180 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI: 180 mg QD oral (PO) lunresertib daily in combination with 180 mg/m2 intravenous (IV) irinotecan given over 30 to 90 minutes, 400 mg/m2 IV leucovorin given over 30 to 90 minutes with irinotecan, and 400 mg/m2 IV fluorouracil bolus after leucovorin, then 2400 mg/m2 IV continuous IV of fluorouracil over 46 hours (Days 1 and 2) of each 14-day cycle
- 240 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI: 240 mg QD oral (PO) lunresertib daily in combination with 180 mg/m2 intravenous (IV) irinotecan given over 30 to 90 minutes, 400 mg/m2 IV leucovorin given over 30 to 90 minutes with irinotecan, and 400 mg/m2 IV fluorouracil bolus after leucovorin, then 2400 mg/m2 IV continuous IV of fluorouracil over 46 hours (Days 1 and 2) of each 14-day cycle
- 60 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI: 60 mg BID oral (PO) lunresertib daily in combination with 180 mg/m2 intravenous (IV) irinotecan given over 30 to 90 minutes, 400 mg/m2 IV leucovorin given over 30 to 90 minutes with irinotecan, and 400 mg/m2 IV fluorouracil bolus after leucovorin, then 2400 mg/m2 IV continuous IV of fluorouracil over 46 hours (Days 1 and 2) of each 14-day cycle
- 80 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI: 80 mg BID oral (PO) lunresertib daily in combination with 180 mg/m2 intravenous (IV) irinotecan given over 30 to 90 minutes, 400 mg/m2 IV leucovorin given over 30 to 90 minutes with irinotecan, and 400 mg/m2 IV fluorouracil bolus after leucovorin, then 2400 mg/m2 IV continuous IV of fluorouracil over 46 hours (Days 1 and 2) of each 14-day cycle
- 80 mg BID RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI: 80 mg BID oral (PO) lunresertib 3 days on and 4 days off in combination with 180 mg/m2 intravenous (IV) irinotecan given over 30 to 90 minutes, 400 mg/m2 IV leucovorin given over 30 to 90 minutes with irinotecan, and 400 mg/m2 IV fluorouracil bolus after leucovorin, then 2400 mg/m2 IV continuous IV of fluorouracil over 46 hours (Days 1 and 2) of each 14-day cycle
- 120 mg QD RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI: 120 mg BID oral (PO) lunresertib 3 days on and 4 days off in combination with 180 mg/m2 intravenous (IV) irinotecan given over 30 to 90 minutes, 400 mg/m2 IV leucovorin given over 30 to 90 minutes with irinotecan, and 400 mg/m2 IV fluorouracil bolus after leucovorin, then 2400 mg/m2 IV continuous IV of fluorouracil over 46 hours (Days 1 and 2) of each 14-day cycle
Period: Overall Study
Arm/Group | 40 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 120 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 180 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 240 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 60 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI | 80 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI | 80 mg BID RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI | 120 mg QD RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI
Started | 2 | 3 | 9 | 4 | 7 | 3 | 4 | 6
Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not Completed | 2 | 3 | 9 | 3 | 7 | 3 | 3 | 5
Not completed — Death | 2 | 3 | 3 | 2 | 2 | 1 | 1 | 3
Not completed — Sponsor Decision to Terminate Study | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0
Not completed — Other Reasons | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 40 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 120 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 180 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 240 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 60 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI | 80 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI | 80 mg BID RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI | 120 mg QD RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI | Total
Number analyzed (Participants) | 2 | 3 | 9 | 4 | 7 | 3 | 4 | 6 | 38
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 51 [49 to 53] | 55 [51 to 59] | 58 [50 to 73] | 66 [55 to 70] | 68 [31 to 75] | 42 [38 to 60] | 44 [41 to 53] | 61 [46 to 78] | 55.5 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 1 | 3 | 3 | 3 | 3 | 17
  Male | 1 | 3 | 6 | 3 | 4 | 0 | 1 | 3 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 0 | 2 | 5 | 3 | 5 | 3 | 3 | 4 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  United States | 2 | 3 | 4 | 1 | 6 | 0 | 2 | 6 | 24
  United Kingdom | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 6
  Spain | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 6
Gene Type [Number; unit: participants]
  CCNE1 | 0 | 0 | 4 | 0 | 2 | 0 | 2 | 4 | 12
  FBXW7 | 2 | 3 | 5 | 4 | 5 | 3 | 2 | 2 | 26

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of RP 6306 in Combination With FOLFIRI
Description: Incidence of grade 3 and above Treatment Related Emergent Adverse Events (TRAEs)
Time Frame: Start of treatment to 30 days post last dose. up to 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 120 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 180 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 240 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 60 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI | 80 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI | 80 mg BID RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI | 120 mg QD RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI
Number analyzed (Participants) | 2 | 3 | 9 | 4 | 7 | 3 | 4 | 6
Participants | 1 | 1 | 6 | 3 | 0 | 1 | 2 | 4

2. Primary Outcome: Recommended Phase 2 Dose (RP2D) and Schedule of RP-6306 in Combination With FOLFIRI
Description: Evaluation of dose-limiting toxicities (DLTs) at or below a frequency of 25%.
Time Frame: During 28 days (2 cycles) from the initiation of the study treatment
Population: DLT evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 120 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 180 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 240 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 60 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI | 80 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI | 80 mg BID RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI | 120 mg QD RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI
Number analyzed (Participants) | 2 | 3 | 5 | 3 | 5 | 2 | 2 | 4
Participants | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Start of treatment to 30 days post last dose. up to 1.5 years
Arm/Group | 40 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 120 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 180 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 240 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI | 60 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI | 80 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI | 80 mg BID RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI | 120 mg QD RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI
All-Cause Mortality (participants affected / at risk) | 2/2 | 3/3 | 3/9 | 2/4 | 2/7 | 1/3 | 1/4 | 3/6
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/3 | 5/9 | 3/4 | 3/7 | 1/3 | 2/4 | 2/6
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 9/9 | 4/4 | 7/7 | 3/3 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI (N=2) | 120 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI (N=3) | 180 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI (N=9) | 240 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI (N=4) | 60 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI (N=7) | 80 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI (N=3) | 80 mg BID RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI (N=4) | 120 mg QD RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Biliary infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium Difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphatamia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Acute Kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI (N=2) | 120 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI (N=3) | 180 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI (N=9) | 240 mg QD RP-6306 (Lunresertib) Daily + FOLFIRI (N=4) | 60 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI (N=7) | 80 mg BID RP-6306 (Lunresertib) Daily + FOLFIRI (N=3) | 80 mg BID RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI (N=4) | 120 mg QD RP-6306 (Lunresertib) 3 Days on and 4 Days Off + FOLFIRI (N=6)
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 3 | 2 | 0 | 0 | 2 | 4
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 1 | 1 | 0 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dry Eye (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 5 | 2 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 3 | 3 | 0 | 2 | 4
Vomitting (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 3 | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 4 | 2 | 0 | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 4 | 1 | 5 | 1 | 1 | 3
Mucosal inflammation (General disorders) | 1 | 2 | 2 | 2 | 2 | 2 | 1 | 3
Pyrexia (General disorders) | 1 | 1 | 4 | 1 | 1 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 2
Candida infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
SAR-COV-2 test positive (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 3 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Hyponatramia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 2
Taste Disorder (Nervous system disorders) | 2 | 2 | 0 | 1 | 2 | 0 | 0 | 0
dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1
dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Reproductive system and breast disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 0 | 2 | 0 | 0 | 3
rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 2 | 0 | 0 | 2
palmar-plantar Erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
skin discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT05147350/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT05147350/SAP_001.pdf